CLINICAL TRIAL: NCT00291499
Title: Clinical Evaluation of Condrosulf 800 mg in the Treatment of Symptomatic OA of the Hand: a 6-month, Double-blind, Placebo Controlled Study
Brief Title: Efficacy Study of Condrosulf in the Treatment of Symptomatic OA of the Hand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03CH/Ct06
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthrosis
Keywords: symptomatic OA of the hand
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Chondroitin 4&6 sulfate (Condrosulf) (Active Comparator)
  Interventions: Drug: Chondroitin 4&6 sulfate (Condrosulf)
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Chondroitin 4&6 sulfate (Condrosulf) — 800 mg/day for 6 months
  Arms: Chondroitin 4&6 sulfate (Condrosulf)
Other: Placebo — 800 mg placebo/day for 6 months
  Arms: placebo

SUMMARY:
The goal of the present study is to investigate the effectiveness of Condrosulf® 800 mg tablets vs. placebo once a day for 6 months in the symptomatic treatment of finger joint osteoarthritis.

Primary endpoints of the study are the evaluation of global spontaneous pain (Huskisson's Visual Analogue Scale: VAS) and the score of Dreiser's algo-functional index (FIHOA) during the treatment with the tested product, Condrosulf®, versus placebo.

DETAILED DESCRIPTION:
The goal of the present study is to investigate the effectiveness of Condrosulf® 800 mg tablets vs. placebo once a day for 6 months in the symptomatic treatment of finger joint osteoarthritis in 160 randomised patients.

Primary endpoints:

Primary endpoints of the study are the evaluation of global spontaneous pain (Huskisson's Visual Analogue Scale: VAS) and the score of Dreiser's algo-functional index (FIHOA) during the treatment with the tested product, Condrosulf®, versus placebo.

Secondary endpoints are:

Efficacy evaluation: Global impression of efficacy expressed by the patient and the physician (VAS), Grip strength (measured manometrically); Morning stiffness duration; Consumption of Paracetamol; Tolerability (4-point verbal scale); Adverse Events occurring during the treatment period; Other parameters:Treatment compliance; Biological markers of arthritis

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex
* Aged 40 and over
* Outpatients
* Patients fulfilling the American Congress of Rheumatology (ACR) criteria for the reporting of hand OA
* Patients showing X-ray features of hand OA on at least two joints (2 IP and/or 1 IP and 1 TMC) of the dominant hand on standard plain radiographs (< 6 month).
* Suffering from regular spontaneous pain on the dominant hand (VAS > or = 40 mm at inclusion time).
* Showing a FIHOA score > or = 6.
* Having had at least two painful flares in a finger joint during the previous 12 month.
* Patients who have signed the written informed consent for their participation in the study
* Patients able to understand and follow the protocol.
* Patients with a satisfying health and nutritional status.
* Female subjects of childbearing potential using, within three months prior to the inclusion in the study, a reliable form of contraception during the course of the study (oral contraceptive pill, intrauterine device or condoms) or female of non childbearing potential (hysterectomy, bilateral ovariectomy or tubal section/ligation).
* Female subjects of childbearing potential with a negative urinary pregnancy test before the inclusion in the study.

Exclusion Criteria:

* Inflammatory joint disease of other origin
* Septic arthritis
* Chronic inflammatory joint disease
* Previous articular fracture of the concerned articulations
* Use of analgesic therapy for other indications
* Receiving oral corticosteroids
* Mono-articular posttraumatic OA of the finger
* Planning surgery of the hands in the following 6 months
* Patients suffering or having suffered from secondary osteoarthritis after one of the following diseases:

  * Infectious arthritis - Acromegaly
  * Ochronosis - Hemachromatosis
  * Gout - Wilson's disease
  * Chondrocalcinosis - Paget's disease
  * Osteochondrosis - Mutation of collagen
  * Genetic problems (for ex. hypermobility) - Previous joint fracture
  * Arthropathies of different aetiologies - Algodystrophy (M. Sudeck)
* Congenital abnormalities
* Recurrent pseudogout
* Major dysplasias
* Intra-articular injection in a hand joint from less than 3 months
* Basic treatment of arthritis with symptom-modifying agents (chondroitin sulfate, glucosamine sulfate, diacerhein, hyaluronic acid) in the last 3 months
* Articular lavage in the last 3 months
* Treatment with corticoids, by any administration route during the last month
* Patient suffering from frequent asthma crises
* Physiotherapy, re-education, alternative medicine (mesotherapy, acupuncture) on the hands foreseeable in the next year
* Serious organic diseases: heart failure, renal or hepatic insufficiency, blood dyscrasia, serious infection
* Participation in other clinical trials in the two months preceding the study
* Known or ascertained hypersensitivity to the active ingredient of the tested drug.
* Patients refusing to sign the written informed consent form
* Patients who do not co-operate, not respecting the protocol requirements
* Pregnant or lactating women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cem Gabay, Prof. Dr., Principal Investigator — HUG - Hôpitaux universitaires de Genève

REFERENCES:
- [Background] Lequesne M. [Symptomatic slow-action anti-arthritic agents: a new therapeutic concept?]. Rev Rhum Ed Fr. 1994 Feb;61(2):75-9. No abstract available. French. PMID 7920505
- [Background] Michel BA, Stucki G, Frey D, De Vathaire F, Vignon E, Bruehlmann P, Uebelhart D. Chondroitins 4 and 6 sulfate in osteoarthritis of the knee: a randomized, controlled trial. Arthritis Rheum. 2005 Mar;52(3):779-86. doi: 10.1002/art.20867. PMID 15751094
- [Background] Uebelhart D, Malaise M, Marcolongo R, de Vathaire F, Piperno M, Mailleux E, Fioravanti A, Matoso L, Vignon E. Intermittent treatment of knee osteoarthritis with oral chondroitin sulfate: a one-year, randomized, double-blind, multicenter study versus placebo. Osteoarthritis Cartilage. 2004 Apr;12(4):269-76. doi: 10.1016/j.joca.2004.01.004. PMID 15023378
- [Background] Cicuttini FM, Spector TD. Osteoarthritis in the aged. Epidemiological issues and optimal management. Drugs Aging. 1995 May;6(5):409-20. doi: 10.2165/00002512-199506050-00007. PMID 7647428
- [Background] Howell DS, Altman RD. Cartilage repair and conservation in osteoarthritis. A brief review of some experimental approaches to chondroprotection. Rheum Dis Clin North Am. 1993 Aug;19(3):713-24. PMID 8210583
- [Background] Volpi N. Oral bioavailability of chondroitin sulfate (Condrosulf) and its constituents in healthy male volunteers. Osteoarthritis Cartilage. 2002 Oct;10(10):768-77. doi: 10.1053/joca.2002.0824. PMID 12359162
- [Background] Conte A, de Bernardi M, Palmieri L, Lualdi P, Mautone G, Ronca G. Metabolic fate of exogenous chondroitin sulfate in man. Arzneimittelforschung. 1991 Jul;41(7):768-72. PMID 1772467
- [Background] Morreale P, Manopulo R, Galati M, Boccanera L, Saponati G, Bocchi L. Comparison of the antiinflammatory efficacy of chondroitin sulfate and diclofenac sodium in patients with knee osteoarthritis. J Rheumatol. 1996 Aug;23(8):1385-91. PMID 8856618
- [Background] Ronca F, Palmieri L, Panicucci P, Ronca G. Anti-inflammatory activity of chondroitin sulfate. Osteoarthritis Cartilage. 1998 May;6 Suppl A:14-21. doi: 10.1016/s1063-4584(98)80006-x. PMID 9743814
- [Background] Uebelhart D, Thonar EJ, Zhang J, Williams JM. Protective effect of exogenous chondroitin 4,6-sulfate in the acute degradation of articular cartilage in the rabbit. Osteoarthritis Cartilage. 1998 May;6 Suppl A:6-13. doi: 10.1016/s1063-4584(98)80005-8. PMID 9743813
- [Background] Bourgeois P, Chales G, Dehais J, Delcambre B, Kuntz JL, Rozenberg S. Efficacy and tolerability of chondroitin sulfate 1200 mg/day vs chondroitin sulfate 3 x 400 mg/day vs placebo. Osteoarthritis Cartilage. 1998 May;6 Suppl A:25-30. doi: 10.1016/s1063-4584(98)80008-3. PMID 9743816
- [Background] Mazieres B, Loyau G, Menkes CJ, Valat JP, Dreiser RL, Charlot J, Masounabe-Puyanne A. [Chondroitin sulfate in the treatment of gonarthrosis and coxarthrosis. 5-months result of a multicenter double-blind controlled prospective study using placebo]. Rev Rhum Mal Osteoartic. 1992 Jul-Sep;59(7-8):466-72. French. PMID 1485136
- [Background] Bucsi L, Poor G. Efficacy and tolerability of oral chondroitin sulfate as a symptomatic slow-acting drug for osteoarthritis (SYSADOA) in the treatment of knee osteoarthritis. Osteoarthritis Cartilage. 1998 May;6 Suppl A:31-6. doi: 10.1016/s1063-4584(98)80009-5. PMID 9743817
- [Background] Uebelhart D, Thonar EJ, Delmas PD, Chantraine A, Vignon E. Effects of oral chondroitin sulfate on the progression of knee osteoarthritis: a pilot study. Osteoarthritis Cartilage. 1998 May;6 Suppl A:39-46. doi: 10.1016/s1063-4584(98)80011-3. PMID 9743819
- [Background] Verbruggen G, Goemaere S, Veys EM. Chondroitin sulfate: S/DMOAD (structure/disease modifying anti-osteoarthritis drug) in the treatment of finger joint OA. Osteoarthritis Cartilage. 1998 May;6 Suppl A:37-8. doi: 10.1016/s1063-4584(98)80010-1. PMID 9743818
- [Background] Verbruggen G, Goemaere S, Veys EM. Systems to assess the progression of finger joint osteoarthritis and the effects of disease modifying osteoarthritis drugs. Clin Rheumatol. 2002 Jun;21(3):231-43. doi: 10.1007/s10067-002-8290-7. PMID 12111630
- [Background] Dreiser RL, Maheu E, Guillou GB, Caspard H, Grouin JM. Validation of an algofunctional index for osteoarthritis of the hand. Rev Rhum Engl Ed. 1995 Jun;62(6 Suppl 1):43S-53S. PMID 7583182
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Gray R, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hand. Arthritis Rheum. 1990 Nov;33(11):1601-10. doi: 10.1002/art.1780331101. PMID 2242058
- [Derived] Gabay C, Medinger-Sadowski C, Gascon D, Kolo F, Finckh A. Symptomatic effects of chondroitin 4 and chondroitin 6 sulfate on hand osteoarthritis: a randomized, double-blind, placebo-controlled clinical trial at a single center. Arthritis Rheum. 2011 Nov;63(11):3383-91. doi: 10.1002/art.30574. PMID 21898340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Started | 81 | 82
Intention to Treat (ITT) | 80 | 82
Per Protocol (PP) | 72 | 67
Safety Population | 81 | 82
Completed | 72 | 67
Not Completed | 9 | 15
Not completed — Adverse Event | 3 | 8
Not completed — Change to other therapy | 2 | 1
Not completed — Intercurrent illness | 1 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Other reasons | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] — Years
  years | 63.9 (8.5) | 63.0 (7.2) | 63.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 62 | 120
  Male | 22 | 20 | 42
Region of Enrollment [Number; unit: participants] — Switzerland
  participants
    Switzerland | 80 | 82 | 162
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (4.5) | 25.0 (3.8) | 25.9 (4.2)
Handedness (no. with dominant left/right hand) [Number; unit: participants] — Number of patients with dominant left hand / dominant right hand
  participants
    left hand | 25 | 26 | 51
    right hand | 55 | 56 | 111
Handedness (no. with target left/right hand) [Number; unit: participants] — Number of patients with target (more painful) left hand / target (more painful) right hand
  participants
    left hand | 23 | 27 | 50
    right hand | 57 | 55 | 112
Symptom duration, mean +/- SD (standard deviation) years, left/right hand [Mean (Standard Deviation); unit: years]
  left hand | 6.9 (6.3) | 6.2 (5.3) | 6.5 (5.8)
  right hand | 7.1 (6.1) | 6.7 (5.7) | 6.9 (5.9)
No. of painful flares in 12 months, mean +/- SD (standard deviation) [Mean (Standard Deviation); unit: flares] | 35.2 (80.0) | 30.0 (70.3) | 32.6 (75.1)
No. of proximal interphalangeal (PIP) nodal joints, mean +/- SD (standard deviation) left/right hand [Mean (Standard Deviation); unit: number of joints]
  left hand | 1.0 (1.5) | 0.9 (1.2) | 0.9 (1.3)
  right hand | 1.2 (1.6) | 1.0 (1.2) | 1.0 (1.4)
No. distal interphalangeal (DIP) nodal joints, mean +/- SD (standard deviation), left/right hand [Mean (Standard Deviation); unit: number of joints]
  left hand | 2.1 (1.4) | 2.0 (1.4) | 2.1 (1.4)
  right hand | 2.4 (1.3) | 2.1 (1.4) | 2.2 (1.3)
Patient's assess. of global hand pain, mean +/- SD (standard deviation), left/right/target hand [Mean (Standard Deviation); unit: mm] — Pain measured with a Visual Analogue Scale (0-100mm where 0=no pain, 100=maximum pain)
  mm
    left hand | 43.8 (21.0) | 42.4 (21.4) | 43.1 (21.2)
    right hand | 48.7 (19.3) | 45.9 (19.2) | 47.3 (19.2)
    target hand | 54.9 (14.2) | 53.6 (14.2) | 54.2 (14.2)
Functional Index for Hand Osteoarthritis (FIHOA) score, mean +/- SD (standard deviation) [Mean (Standard Deviation); unit: units on a scale] — Functional Index for Hand Osteoarthritis (Dreiser's Index). Range 0-30 Patients reported the severity of their symptoms by answering a set of 10 questions. Severity was rated on a numerical scale (0 = possible without difficulty, 1 = possible with slight difficulty, 2 =possible with great difficulty, and 3 = impossible), being 30 points the worst possible pain score
  units on a scale | 11.0 (4.2) | 10.3 (3.8) | 10.7 (4)
No. of fingers with osteophytes on PIP joints, mean +/- SD (standard deviation), left/right hand [Mean (Standard Deviation); unit: number of fingers]
  left hand | 1.9 (1.6) | 1.9 (1.5) | 1.9 (1.6)
  right hand | 2.3 (1.5) | 1.9 (1.5) | 2.1 (1.5)
No. of fingers with osteophytes on DIP joints, mean +/- SD (standard deviation), left/right hand [Mean (Standard Deviation); unit: number of fingers]
  left hand | 2.9 (1.3) | 3.0 (1.2) | 3.0 (1.2)
  right hand | 3.1 (1.3) | 3.1 (1.1) | 3.1 (1.2)
No. of patients with erosive hand OA [Number; unit: participants] | 26 | 35 | 61
No. of patients with rhizarthrosis [Number; unit: participants] | 37 | 43 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Spontaneous Pain Intensity of Target Hand
Description: Intensity of global spontaneous pain is evaluated by the patient himself on a Huskisson's visual analogue scale (VAS) of 100 mm. 0=no pain 100=max pain Change calculated as difference between Month 6 value and baseline value target hand is defined as the patient's most symptomatic hand or, when both hands were equally painful, the patient's dominant hand.
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Number analyzed (Participants) | 80 | 82
mm | -20 (26) | -11.3 (24)
Statistical Analysis 1: Comparison: Chondroitin 4&6 Sulfate (Condrosulf) vs Placebo; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -8.7

2. Primary Outcome: Change in Functional Index for Hand Osteoarthritis Dreiser's Score (FIHOA) in the Target Hand
Description: Functional Index for Hand Osteoarthritis (Dreiser's Index). Range 0-30 Patients reported the severity of their symptoms by answering a set of 10 questions. Severity was rated on a numerical scale (0 = possible without difficulty, 1 = possible with slight difficulty, 2 =possible with great difficulty, and 3 = impossible), being 30 points the worst possible pain score.
  Change calculated as difference between the month 6 value and baseline value
  Target hand defined as the patient's most symptomatic hand or, when both hands were equally painful, the patient's dominant hand
Time Frame: 6 month
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Number analyzed (Participants) | 80 | 82
score on a scale | -2.9 (5.3) | -0.7 (4.8)
Statistical Analysis 1: Comparison: Chondroitin 4&6 Sulfate (Condrosulf) vs Placebo; Test type: Superiority; p = 0.008, t-test, 2 sided; Mean Difference (Final Values) = -2.14

3. Secondary Outcome: Investigator Global Evaluation on Efficacy
Description: Global impression of the efficacy judged by the Investigators at month 6 by means of a visual analogue scale from 0 (no efficacy) to 100 mm (very good efficacy)
Time Frame: 6 months
Population: ITT (missing values where not replaced)
Measure: Count of Participants; unit: Participants
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Number analyzed (Participants) | 79 | 76
Participants
  marked improvement of the clinical condition | 15 | 9
  slight improvement of the clinical condition | 20 | 16
  doubtful improvement of the clinical condition | 16 | 10
  no improvement | 28 | 41
Statistical Analysis 1: Comparison: Chondroitin 4&6 Sulfate (Condrosulf) vs Placebo; Test type: Superiority; p = 0.043, Cochran-Mantel-Haenszel — Threshold p <0.05

4. Secondary Outcome: Change in Grip Strength
Description: Grip strength determined on both hands using a Jamar dynamometer.Patients were required to grip the dynamometer handle and squeeze as hard as possible according to their individual pain limits. The right hand grip was measured first, then the left; this procedure was performed 3 times. The mean value of these 3 measurements was recorded.
  Change calculated as difference between the month 6 value and baseline value
Time Frame: 6 months
Population: ITT (missing values were not replaced)
Measure: Mean (Standard Deviation); unit: Kg/cm^2
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Number analyzed (Participants) | 70 | 68
Kg/cm^2 | 2.5 (6.6) | 0.6 (5.8)
Statistical Analysis 1: Comparison: Chondroitin 4&6 Sulfate (Condrosulf) vs Placebo; Test type: Superiority; p = 0.132, Wilcoxon (Mann-Whitney) — Threshold p<0.05

5. Secondary Outcome: Change in Morning Stiffness Duration
Description: Change in morning stiffness duration calculated as the difference between the month 6 value and the baseline value
Time Frame: 6 months
Population: ITT (missing values were not replaced)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Number analyzed (Participants) | 72 | 67
minutes | -4.8 (16.6) | 0.3 (12.0)
Statistical Analysis 1: Comparison: Chondroitin 4&6 Sulfate (Condrosulf) vs Placebo; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney) — Threshold p<0.05

6. Secondary Outcome: Consumption of Paracetamol
Description: Total consumption (between ^baseline and month 6) of paracetamol (500 mg tablets) reported by the patients on a daily diary
Time Frame: 6 months
Population: ITT (missing values were not replaced)
Measure: Mean (Standard Deviation); unit: tablets/week
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
Number analyzed (Participants) | 78 | 76
tablets/week | 1.9 (2.8) | 2.0 (4.2)
Statistical Analysis 1: Comparison: Chondroitin 4&6 Sulfate (Condrosulf) vs Placebo; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.363

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Chondroitin 4&6 Sulfate (Condrosulf) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 2/81 | 2/82
Other Adverse Events (participants affected / at risk) | 5/81 | 4/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chondroitin 4&6 Sulfate (Condrosulf) (N=81) | Placebo (N=82)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
synus tachicardia (Cardiac disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chondroitin 4&6 Sulfate (Condrosulf) (N=81) | Placebo (N=82)
Diarrhea (Gastrointestinal disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No